CLINICAL TRIAL: NCT03836781
Title: Comparison of Teh TEMPEffect of Subgingival Irrigation Wif Ketorolac and Chlorhexidine in Patients Wif Chronic Periodontist.
Brief Title: Teh Effect of Subgingival Irrigation Wif Ketorolac and Chlorhexidine in Patients Wif Chronic Periodontist
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Amirhossein Farahmand (Other)
Responsible Party: Sponsor-Investigator, Amirhossein Farahmand, assistant prof, Islamic Azad University, Sanandaj
Organization: Islamic Azad University, Sanandaj (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2037
Record Dates: First submitted 2019-02-08; First posted 2019-02-11 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Ketorolac

STUDY DESIGN:
Intervention Model Description: split mouth
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketorolac 3% (Active Comparator): ketorolac 3% topical subgingival irrigation was put into the periodontal pocket using an insulin syringe
  Interventions: Drug: Ketorolac
- chlorhexidine 2% (Other): chlorhexidine 2% topical subgingival irrigation was put into the periodontal pocket using an insulin syringe
  Interventions: Drug: Chlorhexidine 2%

INTERVENTIONS:
Drug: Ketorolac — Ketorolac 3% topical subgingival irrigation was put into the periodontal pocket using an insulin syringe
  Other Names: Group A
  Arms: ketorolac 3%
Drug: Chlorhexidine 2% — Chlorhexidine 2% topical subgingival irrigation was put into the periodontal pocket using an insulin syringe
  Other Names: Group B
  Arms: chlorhexidine 2%

SUMMARY:
In this study, 40 patients with a history of Mild- Periodontitis who were diagnosed with clinical and radiographic findings showed that all of the periodontal parameters before the treatment, during the treatment period Then, scaling & Root planing and oral hygiene instructions were given to the patients, and after 2 weeks, the patients who received the study were randomly divided into two groups (Balanced Block Randomization) with four blocks according to the visit time. To group A, oral chlorohexidine and to B group, the drug Ketorolac was given. 5 mm of the drugs required every 15 days the areas underwent a gingival wash with an insulin syringe, which lasted for 3 months.

DETAILED DESCRIPTION:
In this study, 40 patients with a history of Mild- Periodontitis who were diagnosed with clinical and radiographic findings showed that all of the periodontal parameters before the treatment, during the treatment period Then, scaling & Root planing and oral hygiene instructions were given to the patients, and after 2 weeks, the patients who received the study were randomly divided into two groups (Balanced Block Randomization) with four blocks according to the visit time. To group A, oral chlorohexidine (Ghol Darou-Tehran) and to B group, the drug Ketorolac (Exir-Boroujerd) was given. 5 mm of the drugs required every 15 days the areas underwent a gingival wash with an insulin syringe, which lasted for 3 months. Pl, BI, PD were evaluated in the study sessions. At the end of the clinical change, a multiple measure ANOVA test was used to compare the preceding and follow-up sessions in both groups, considering the intervention method as Between subject comparison And measured at the time of measurement as a Repeated Factor.

ELIGIBILITY:
Inclusion Criteria:

40 patients with periodontitis chronic and has a 2 molar symmetrically in the lower jaw pockets of the periodontal depth of at least 5 mm and CAL 1-2 mm in at least one of the surfaces of the teeth, were selected

Exclusion Criteria:

1. systemic disease
2. pregnancy or breastfeeding
3. allergy drug used
4. smoking
5. medication 6. not willing to consent to participate in the study

7-Trismus 8-The type of disease periodontal (Aggressive) 9. History of periodontal treatment in the previous 6 months 10-orthodontic treatment

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2019-06-08 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Pocket depth | 3 month
  Clinical periodontal measurements to Williams periodontal probe

CONTACTS AND LOCATIONS:
Locations (1):
- Amirhossein Farahmand, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No